CLINICAL TRIAL: NCT01023295
Title: OXiGENE OXC402-201: A Phase 2, Randomized, Double-Masked, Placebo-Controlled Study of the Safety, Pharmacokinetics, and Biological Effects of Intravenous Fosbretabulin in Asian Subjects With Polypoidal Choroidal Vasculopathy (PCV)
Brief Title: Study Evaluating the Safety and Response of Fosbretabulin in Asian Patients With Polypoidal Choroidal Vasculopathy (PCV)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mateon Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OXC402-201
Record Dates: First submitted 2009-11-30; First posted 2009-12-02 (Estimated); Last update posted 2011-11-01 (Estimated); Status verified 2011-10

CONDITIONS: Polypoidal Choroidal Vasculopathy
Keywords: Polypoidal Choroidal Vasculopathy; PCV; Polypoid; oxigene; VDA; vascular disrupting agent; combretastatin; fosbretabulin
MeSH Terms: conditions — Polypoidal Choroidal Vasculopathy | interventions — fosbretabulin; combretastatin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Placebo (Placebo Comparator): single dose
  Interventions: Drug: Saline
- 15 mg/m^2 (Experimental): 15 mg/m^2 fosbretabulin, single dose
  Interventions: Drug: fosbretabulin
- 25 mg/m^2 (Experimental): 25 mg/m^2 fosbretabulin, single dose
  Interventions: Drug: fosbretabulin
- 35 mg/m^2 (Experimental): 35 mg/m^2 fosbretabulin, single dose
  Interventions: Drug: fosbretabulin
- 45 mg/m^2 (Experimental): 45 mg/m^2 fosbretabulin, single dose
  Interventions: Drug: fosbretabulin

INTERVENTIONS:
Drug: fosbretabulin — single dose, intravenous infusion
  Other Names: combretastatin; CA4P
  Arms: 15 mg/m^2; 25 mg/m^2; 35 mg/m^2; 45 mg/m^2
Drug: Saline — single dose, intravenous infusion
  Arms: Placebo

SUMMARY:
The primary objective of this study is to examine effects of fosbretabulin tromethamine (fosbretabulin) on PCV as reflected by a change from baseline in the number of polypoid lesions on indocyanine green angiography (ICGA).

ELIGIBILITY:
Inclusion Criteria

* Male or female age ≥21 years.
* Asian race (e.g. Chinese, Japanese, Korean, Thai).
* Polypoidal choroidal vasculopathy in the study eye
* Presence of ≥ 1 visible polypoidal varicosity on ICGA.
* Presence of a measurable branching vascular network
* BCVA by ETDRS of 68 to 4 letters in the study eye.

Ophthalmologic Exclusion Criteria

* Prior treatment with intravitreal or systemic anti-VEGF therapy within 60 days of enrollment.
* Any other prior treatment for PCV including thermal laser photocoagulation, photodynamic therapy (i.e., verteporfin), or any investigational therapies.
* Any history of prior retinal or subretinal surgery, transpupillary thermography, radiation, implantation of intravitreal drug delivery device, vitrectomy.
* Any other intraocular surgery or laser treatment within 90 days or any surgeries planned during the study period.
* Fibrosis involving ≥50% of the total lesion.
* Presence of hemorrhage which potentially obscures >75% of vascular pathology to be assessed by imaging procedures.
* Retinal or choroidal vascular disease in study eye due to causes other than PCV, such as uveitis, trauma, or pathologic myopia.
* Macular edema in either eye due to other causes, such as diabetic retinopathy.
* Evidence of glaucomatous eye disease, glaucomatous visual field loss.
* History of allergy to fluorescein or ICG dye.

Medical Exclusion Criteria

* Current or history within two years of any significant heart disease.
* Uncontrolled hypertension.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-07; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Evaluate change in number of polypoid lesions on ICGA from baseline to Day 2 | from baseline to Day 2
Evaluate change in the number of polypoid lesions on ICGA from baseline to Day 8 | from baseline to Day 8

SECONDARY OUTCOMES:
Evaluate the change in area of the branching vascular network of PCV using ICGA from baseline to Day 2 | baseline to Day 2
Evaluate the change in the area of branching vascular network of PCV on ICGA from baseline to Day 8 | baseline to Day 8
Examine effects of fosbretabulin on choroidal neovasculariztion (CNV) and total lesion size using fluorescein angiography (FA) | Day 29

CONTACTS AND LOCATIONS:
Locations (5):
- OXiGENE Investigational Site, Los Angeles, California, United States
- OXiGENE Investigational Site, Hong Kong, Hong Kong
- OXiGENE Investigational Site, Singapore, Singapore
- OXiGENE Investigational Site, Seoul, South Korea
- OXiGENE Investigational Site, Changhua, Taiwan